CLINICAL TRIAL: NCT01096329
Title: A Phase 1, Open-label, Randomized, Three-cohort, Two-period Crossover Study to Determine the Relative Bioavailability of Testosterone Following Application of Two Testosterone Transdermal Spray (TTS) Formulations Once Daily and Intrinsa® Patch Twice Weekly in Healthy, Surgically and Naturally Post-menopausal Women Receiving Estrogen Replacement Therapy
Brief Title: A Pharmacokinetic (PK) Study to Compare the Absorption of Two Formulations of Transdermal Testosterone Spray and Intrinsa®
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wes Day, PhD/VP Clinical, Vivus Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: VTS-102
Record Dates: First submitted 2010-03-28; First posted 2010-03-31 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: postmenopausal; hormone replacement therapy
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 2 (Active Comparator): Testosterone Spray (5%) vs Intrinsa® Patch
  Interventions: Drug: Intrinsa® Patch and Testosterone Spray 5%
- Cohort 3 (Active Comparator): Testosterone Spray (1%) vs Intrinsa® Patch
  Interventions: Drug: Intrinsa® Patch and Testosterone Spray 1%
- Cohort 1 (Active Comparator): Testosterone Spray (5%) vs Testosterone Spray (1%)
  Interventions: Drug: Testosterone Spray 5% and 1%

INTERVENTIONS:
Drug: Testosterone Spray 5% and 1% — Testosterone Spray 5% 2x90uL for 14 days Testosterone Spray 1% 2x90uL for 14 days
  Arms: Cohort 1
Drug: Intrinsa® Patch and Testosterone Spray 5% — Testosterone Spray 5% 2x90uL for 14 days Intrinsa® Patch for 14 days
  Arms: Cohort 2
Drug: Intrinsa® Patch and Testosterone Spray 1% — Testosterone Spray 1% 2x90uL for 14 days Intrinsa® Patch for 14 days
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to determine if the absorption of the testosterone spray is the same as the Intrinsa® Patch.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent
2. Naturally or surgically postmenopausal females, 45 - 65 years of age
3. Subjects have spontaneous amenorrhea for at least 12 months
4. Subjects have a serum total testosterone level of < 30 ng/dL
5. Subjects currently on a stable dose of prescribed oral or transdermal estrogen replacement therapy (ERT) for a period of at least 8 to 12 weeks prior to screening, respectively, or not on ERT.
6. A body weight of at least 50 kg and a body mass index (BMI) between 18 and 35 kg/m2, inclusive [BMI will be calculated as weight in kg/(height in m)2]
7. Medically healthy, with clinically insignificant screening results (e.g., laboratory profiles, medical histories, ECGs, physical examination (including breast examination), in the opinion of the Investigator.
8. Subjects are able to communicate with the Investigator, and to understand and to comply with all requirements of study participation.
9. An adequate washout period prior to obtaining any baseline assessments in women who have been previously treated for postmenopausal symptoms. Calculated from study Day 1, the minimum washout period will be 2 and 4 weeks for prior treatment with testosterone oral and transdermal products, respectively, 3 months for prior treatment with testosterone implants and 2 weeks for treatment with estratest.

Exclusion Criteria:

1. A positive serum pregnancy test at screening
2. A history or presence of significant cardiovascular, neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the transdermal absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the Investigator
3. Any clinically significant laboratory abnormalities as judged by the Investigator
4. Subjects are experiencing > 20 hot flushes per week
5. Subjects are suffering from severe acne, moderate to severe hirsutism or androgenic alopecia, or have a history of severe dermatological problems or drug-induced contact dermatitis
6. Systolic blood pressure > 150 mm Hg or diastolic blood pressure > 95 mm Hg at screening or prior to the first dosing in this study (two rechecks are allowed)
7. Any malignancy except basal cell carcinoma
8. A significant psychiatric disorder (e.g., major depression, etc.) that might, in the Investigator's opinion, prevent the subject from completing the study
9. Currently smoke more than 10 cigarettes a day
10. A history of breast biopsy with atypical hyperplasia
11. A prior history of breast cancer, suspected breast cancer, or other current or prior cancer within the past 10 years
12. Exhibits anemia, defined as a hemoglobin level at screening below the laboratory's lower limit of normal reference range
13. Diabetes mellitus
14. Any chronic skin disorder (e.g., eczema, psoriasis) likely to interfere with transdermal drug absorption or assessments of skin tolerability
15. Positive urine drug test and/or positive breath alcohol test at screening or prior to the first dosing in this study (Period 1 only)
16. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV) at screening
17. Any history or presence of alcoholism or drug or substance abuse as defined by the Investigator
18. A history of hypersensitivity or idiosyncratic reaction to testosterone, octisalate, PEG 200, IPA, or other sunscreens, or alcohol-based skin products or Intrinsa®
19. Use of any prescription (except estrogen replacement therapy) or over-the-counter (OTC) medication, within the 30 days prior to the first dosing in this study. Up to 2 g per day of acetaminophen is allowed at the discretion of the Investigator
20. Use of any drugs known to have clinical significance in inhibiting or inducing liver enzymes involved in drug metabolism [CYP P450]) within 30 days prior to the first dosing in this study. Use of any systemic corticosteroids within 30 days prior to the first dosing in this study
21. Blood donation or significant blood loss within 56 days prior to the first dosing in this study. Any contraindication to blood sampling
22. Plasma donation within 7 days prior to the first dosing in this study
23. Currently using or has a history of any androgen use within 6 months prior to screening, or uses dehydroepiandrosterone (DHEA) >/= 25 mg per day, or St. John's Wort within 4 weeks prior to baseline. Due to large number of herbal remedies available, all other herbal supplements will be reviewed by the Sponsor during screening
24. Currently using estratest (esterified estrogens and methyltestosterone)
25. Use of an investigational drug within 30 days or six half-lives, whichever is longer, prior to the first dosing in this study
26. Clinical judgment by the Investigator that the subject should not participate in the study
27. Involvement in the planning and conduct of the study (applies to both VIVUS and designee staff, and staff at the investigational site)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To measure the amount of testosterone in the blood after dosing | 2 months
  The following PK parameters of testosterone will be measured AUC0-24, AUC0-48, AUC0-72, AUC0-96, Cavg, Cmin, Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Mark Allison, MD, Principal Investigator — MDS Pharma Services Inc
Locations (1):
- MDS Pharma Services, Tempe, Arizona, United States